CLINICAL TRIAL: NCT01613638
Title: Congenital Malformations and Intrauterine Pollutants Exposure (Alcohol, Solvents and Pesticides) in Brittany. Population Based Case-control Study Short Title : Malformations and Environment Acronym : PENEW for "Pregnancy Environment and Newborn Malformations"
Brief Title: Pregnancy Environment and Newborn Malformations
Acronym: PENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHRC/10-02 - PENEW; B110827-40 (Other: AFSSAPS); 11/22-811 (Other: CPP Ouest V (Rennes)); 2010-A01445-34 (Other: AFSSAPS)
Record Dates: First submitted 2012-05-24; First posted 2012-06-07 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Congenital Malformation
Keywords: congenital malformation; pollutants
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Congenital malformations (Other): All livebirths, fetal deaths with gestational age (GA) ≥22 weeks and terminations of pregnancy (at any gestational age) after prenatal diagnosis of malformation.
  * born from mothers living in Brittany at delivery
  * with a congenital anomaly according to Eurocat criteria, diagnosed or suspected (and then confirmed) at birth
  * or with mild congenital heart defects, genital anomalies or hip dislocation diagnosed after birth (and before the age of one)
  Interventions: Other: meconium samples + maternal self-questionnaire
- control (Other): 2 controls per case will be included, corresponding to the first 2 births without congenital anomalies, with same sex and same birth place, following the case.
  Interventions: Other: meconium samples + maternal self-questionnaire

INTERVENTIONS:
Other: meconium samples + maternal self-questionnaire — meconium samples + maternal self-questionnaire

SUMMARY:
Congenital malformations rate is about 3% in France. There are already 5 registries in France, covering about 16% of French births: Paris Registry, (about 38 000 births /year), Alsace Registry, (about 23 000 births/year), Rhône-Alpes Registry, (about 56 000 births/year), Auvergne Registry, (about 14 000 births/year), and la Réunion Registry. The aim of malformation registries is to carry out epidemiologic surveillance of congenital anomalies. The objectives are mainly to provide essential epidemiologic information on congenital anomalies, to facilitate the early warning of teratogenic exposures, to act as an information and resource centre regarding clusters, to provide data for research related to the causes and prevention of congenital anomalies.

A previous study was carried out in Brittany in 2008-2009, by the perinatal network of Ille et Vilaine, in collaboration with two research teams (Inserm U1085 and Inserm U 936), to record all cases of 4 types of congenital anomalies: congenital heart disease, spina bifida, diaphragmatic hernia and hypospadia. The results showed prevalence rates similar to those observed by Eurocat for spina bifida and diaphragmatic hernia, but a higher prevalence regarding congenital heart diseases and hypospadia. In this study the investigators could not determine whether this was due to a real higher frequency or to a particular exhaustiveness in the recording methodology.

There are hypothesis about the role of intrauterine exposure to pesticides, known as endocrine disruptors, and the risk of congenital genital anomalies. Brittany is an intensive agricultural area, and it is thus worth studying the impact of pesticides exposure on congenital anomalies.

There are also hypothesis on the impact of occupational exposure to solvents on congenital anomalies (Garlantezec 2009), and on the role of alcohol exposure (which concerns about 8% pregnant women in France) on oro-facial clefts and congenital heart diseases.

The Registry of congenital anomalies in Brittany was set up in 2010. The main aim is to study the impact of intra-uterine exposure to solvents, pesticides and alcohol on the risk of congenital malformations diagnosed at births, by measuring the exposure both directly in meconium, and indirectly by questionnaires.

Secondary objectives are to study other risk factors such as medicine intake, pregnancy illness…

DETAILED DESCRIPTION:
Population based case-control study:

2 controls per case will be included, corresponding to the first 2 births without congenital anomalies, with same sex and same birth place, following the case.

INVESTIGATION METHODOLOGY :

All maternity in Brittany were proposed to participate. In each maternity, the referent practitioner informs the parents and includes the cases.

For each case and control, meconium samples and a mother's lock are collected by nurses or midwives, medical data are collected from medical reports by the registry investigator, and a self-questionnaire is filled by the mother.

Meconium samples are immediately stored in a freezer (-20°C), secondarily transported to a biological storage centre at the university hospital and then dispatched to specialised laboratories for toxicological analyses: INERIS (for solvents and pesticides) and Toxicology Unit, University hospital Rennes (for Alcohol).

For dead fetuses (stillbirths or termination of pregnancy), meconium will be collected by the pathologist in charge of the autopsy, after parents' consent.

Evaluation of exposure:

* direct evaluation: by toxicological analyses in meconium samples: Alcohol, Solvents and pesticides
* indirect evaluation: by maternal self-questionnaire including data on occupational and domestic exposures, hobbies, life habits…, precise address (for spatial location)

Particular cases: mild congenital heart defects, genital anomalies and hip dislocation diagnosed later after birth (after the period oh meconium and before the age of one): these cases will be spotted through the Registry, there won't be any biological sample for them, but mothers will be contacted by main investigator and medical data and mother questionnaires will be collected. There won't be any control included for those cases included after birth.

Associations between exposure risk factors (alcohol, solvents and pesticides) and the risk of congenital malformations will be estimated by a multivariate analysis.

* Exposure to solvents will be estimated by assay in meconium and by occupational questionnaire
* Exposure to alcohol will be estimated by assay of Ethylglucuronide et de Ethylsulfate in meconium.
* Exposure to pesticides will be estimated by assay in meconium, by questionnaire and by spatial location.

ELIGIBILITY:
Inclusion Criteria:

All live births, fetal deaths with gestational age (GA) ≥22 weeks and terminations of pregnancy for medical reasons (IMG) from 20 weeks of amenorrhea (SA) included.

* born from mothers living in Brittany at delivery
* with a congenital anomaly according to Eurocat criteria, diagnosed or suspected (and then confirmed) at birth
* or with mild congenital heart defects, genital anomalies or hip dislocation diagnosed after birth (and before the age of one) Suspicion of chromosomal abnormality or genetic syndrome on purely clinical criteria but not yet authenticated by genetic analyzes. If the chromosomal or genetic abnormalities are secondarily authenticated, these cases will be excluded a posteriori.

Non inclusion criteria :

* Spontaneous abortion before 22 weeks gestational age.
* IMG before the 20 week term amenorrhea
* Chromosomal abnormalities or syndromes genetic authenticated by karyotype or analysis in molecular biology, in antenatal
* Mother with legal protection (guardianship)

Exclusion Criteria:

* Prenatally suspected malformations, which are not confirmed by postnatal screening or clinical evolution

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1657 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
impact of intra-uterine exposure to solvents, pesticides and alcohol on the risk of congenital malformations diagnosed at births, by measuring the exposure both directly in meconium, and indirectly by questionnaires. | up to 48 hours
  impact of intra-uterine exposure to solvents, pesticides and alcohol on the risk of congenital malformations diagnosed at births, by measuring the exposure both directly in meconium, and indirectly by questionnaires.

SECONDARY OUTCOMES:
other risk factors such as medicine intake, pregnancy illness… | up to 48 hours
  other risk factors such as medicine intake, pregnancy illness…

CONTACTS AND LOCATIONS:
Overall Officials: Florence Rouget, MD, Principal Investigator — Rennes University Hospital; Philippe Lefevre, MD, Principal Investigator — Fougères Hospital; Joëlle Gueguen, MD, Principal Investigator — Saint-Grégoire Hospital; Isabelle Blanchot, MD, Principal Investigator — Clinique La Sagesse - Rennes; Maria Vernis, MD, Principal Investigator — Saint Malo hospital; Dominique Chaumet, MD, Principal Investigator — Vitré Hospital; Joseph Abi-Fadel, MD, Principal Investigator — Redon Hospital; Philippe Rebour, MD, Principal Investigator — Lannion Hospital; Michel Turban, MD, Principal Investigator — Dinan Hospital; Claire Combescure, MD, Principal Investigator — Saint-Brieuc Hospital; Joseph Magagi, MD, Principal Investigator — Polyclinique du Littoral - Saint-Brieuc; Michel Collet, MD, Principal Investigator — University Hospital, Brest; David Somerville, MD, Principal Investigator — Polyclinique de Keraudren - Brest; Alain Hassoun, MD, Principal Investigator — Clinique Pasteur - Brest; Charles Bellot, MD, Principal Investigator — Quimper Hospital; Philippe Tillaut, MD, Principal Investigator — Lorient Hospital; Hubert Journel, MD, Principal Investigator — Vannes Hospital; Claire Duhaut, MD, Principal Investigator — Clinique Océane - Vannes; Patrick Vallée, MD, Principal Investigator — Pontivy Hospital; Marie-Agnès Guillou, MD, Principal Investigator — Ploermël Hospital
Locations (11):
- France (11):
  - Polyclinique de Keraudren, Brest, Brittany Region
  - Brest University Hospital, Brest, Brittany Region
  - Lannion Hospital, Lannion, Brittany Region
  - Lorient Hospital, Lorient, Brittany Region
  - Ploermel Hospital, Ploërmel, Brittany Region
  - Quimper Hospital, Quimper, Brittany Region
  - Rennes University Hospital, Rennes, Brittany Region
  - Saint-Brieuc Hospital, Saint-Brieuc, Brittany Region
  - Saint-Grégoire Hospital, Saint-Grégoire, Brittany Region
  - Clinique Océane, Vannes, Brittany Region
  - Vannes Hospital, Vannes, Brittany Region

REFERENCES:
- [Background] Meyer-Monath M, Beaumont J, Morel I, Rouget F, Tack K, Lestremau F. Analysis of BTEX and chlorinated solvents in meconium by headspace-solid-phase microextraction gas chromatography coupled with mass spectrometry. Anal Bioanal Chem. 2014 Jul;406(18):4481-90. doi: 10.1007/s00216-014-7836-2. Epub 2014 May 18. PMID 24838489
- [Background] Meyer-Monath M, Chatellier C, Cabooter D, Rouget F, Morel I, Lestremau F. Development of liquid chromatography methods coupled to mass spectrometry for the analysis of substances with a wide variety of polarity in meconium. Talanta. 2015 Jun 1;138:231-239. doi: 10.1016/j.talanta.2015.02.058. Epub 2015 Mar 19. PMID 25863396
- [Background] Meyer-Monath M, Chatellier C, Rouget F, Morel I, Lestremau F. Development of a multi-residue method in a fetal matrix: analysis of meconium. Anal Bioanal Chem. 2014 Dec;406(30):7785-97. doi: 10.1007/s00216-014-8243-4. Epub 2014 Nov 9. PMID 25381610
- [Result] Rouget F, Bihannic A, Cordier S, Multigner L, Meyer-Monath M, Mercier F, Pladys P, Garlantezec R. Petroleum and Chlorinated Solvents in Meconium and the Risk of Hypospadias: A Pilot Study. Front Pediatr. 2021 Jun 2;9:640064. doi: 10.3389/fped.2021.640064. eCollection 2021. PMID 34150682